CLINICAL TRIAL: NCT04342585
Title: Randomised Controlled Trial Comparing Vaginal Pessary and Progestogen as an Intervention in Twin Pregnancy With Short Cervical Length to Prevent Spontaneous Preterm Birth
Brief Title: Comparison Between Vaginal Pessary and Progestogen in Twin Pregnancy With Short Cervical Length
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Rahana Abd Rahman, Co-primary investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JEP-2020-065; DIP-2019-028 (Other Grant/Funding Number: Dana Impak Perdana)
Record Dates: First submitted 2020-04-06; First posted 2020-04-13 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Preterm Birth
Keywords: twin; vaginal pessary; vaginal progestogen; short cervix
MeSH Terms: conditions — Premature Birth | interventions — Utrogestan; Pessaries

STUDY DESIGN:
Intervention Model Description: All women with twin pregnancies will be screened for suitability via measurement of the cervical length at 20 to 24 weeks gestation. Those with a cervical length of 30mm or less will be recruited into the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal progestogen (Active Comparator): 200mg of vaginal progestogen will be inserted before bedtime every day from time of recruitment until 34 weeks gestation.
  Interventions: Drug: Micronised vaginal progesterone
- Vaginal pessary (Active Comparator): Vaginal pessary with an internal diameter size of 32 or 35 mm will be inserted at the time of recruitment and kept until 34 weeks gestation.
  Interventions: Device: Vaginal pessary

INTERVENTIONS:
Drug: Micronised vaginal progesterone — A diary will be given to participants to ensure compliance.
  Other Names: Utrogestan
  Arms: Vaginal progestogen
Device: Vaginal pessary — The internal diameter size will be decided based on the clinical assessment of the cervix.
  Other Names: Arabin pessary
  Arms: Vaginal pessary

SUMMARY:
A randomized clinical trial comparing vaginal progestogen and vaginal pessary as an intervention for twin pregnancies with short cervical length.

DETAILED DESCRIPTION:
This is a randomized controlled trial to compare women with twin pregnancies and diagnosed with asymptomatic short cervical length. Two types of interventions will be compared i.e vaginal progestogen and vaginal pessary.

ELIGIBILITY:
Inclusion Criteria:

* all twin pregnancies
* cervical length less than 30mm

Exclusion Criteria:

* Twin to twin transfusion syndrome
* Stillbirth
* congenital anomaly in one of the fetuses
* previous cervical trauma or surgery
* cervical cerclage in current pregnancy
* premature labour with or without rupture of membranes
* severe vaginal discharge
* acute vaginitis or cervicitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Spontaneous preterm birth | Through study completion up to 37 weeks
  Mean gestational age at delivery in weeks

SECONDARY OUTCOMES:
Maternal age | Pre-intervention
  Mean maternal age in years
Race | Pre-intervention
  Percentage of each race recruited
Maternal body mass index | Pre-intervention
  Mean maternal body mass index in kg/m2 before pregnancy or in the first trimester
Parity | Pre-intervention
  Mean number of parity
Type of twin pregnancy | Pre-intervention
  Chorionicity of twin pregnancy
Type of conception | Pre-intervention
  Method of conception
Gestational age at recruitment | Pre-intervention
  Mean gestational age at recruitment in weeks
Gestational age at commencement of treatment | Pre-intervention
  Mean gestational age at commencement of treatment in weeks
Cervical length before commencement of treatment | Pre-intervention
  Mean cervical length before commencement of treatment in mm
Vaginal infection | Pre-intervention
  Percentage of participants with vaginal infection prior to commencement of treatment
Previous miscarriages | Pre-intervention
  Percentage of participants with previous first and second trimester miscarriages
Pre-existing medical disorders | Pre-intervention
  Percentage of participants with pre-existing medical disorders
Previous spontaneous preterm birth | Pre-intervention
  Percentage of participants with previous spontaneous preterm birth
Antenatal complications | Through study completion up to 37 weeks
  Percentage of participants with antenatal complications
Fetal complications | Through study completion up to 37 weeks
  Percentage of participants with fetal complications
Mode of delivery | Through study completion up to 37 weeks
  Percentage of participants who delivered vaginally or via caesarean section
Intrapartum complications | Throughout labour up to delivery of the neonate
  Percentage of participants with intrapartum complications
Postpartum complications | Through delivery of neonate up to 42 days after delivery
  Percentage of participants with postpartum complications
Total blood loss | Through delivery of neonate up to 42 days after delivery
  Mean total blood loss in ml
Birth weight | Immediately after birth of neonate
  Mean birth weight in grams
Apgar score | Immediately after birth of neonate
  Mean Apgar score
Anthropometry assessment of neonates | Immediately after birth of neonate
  Mean length and head circumference of neonates at birth in cm
Neonatal intensive care unit admission | Immediately after birth of neonate up to discharge (approximately 30 days)
  Percentage of neonates required Neonatal intensive care unit admission
Duration in neonatal intensive care unit | Through neonatal intensive care unit stay up to discharge (approximately 30 days)
  Mean duration in neonatal intensive care unit in days
Neonatal complications | Immediately after birth up to 30 days
  Percentage of neonates with complications

CONTACTS AND LOCATIONS:
Locations (1):
- UKM Medical Centre, Cheras, Kuala Lumpur, Malaysia